CLINICAL TRIAL: NCT00200226
Title: Oral Misoprostol Before Endometrial Biopsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: HIC02.159
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2007-09-21 (Estimated); Status verified 2007-09

CONDITIONS: Endometrial Biopsy
Keywords: pain/discomfort; cervical dilatation; side effects
MeSH Terms: interventions — Misoprostol; Vitamin B 6

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Vitamin B6
  Interventions: Drug: vitamin B6
- 2 (Active Comparator): misoprostol
  Interventions: Drug: misoprostol

INTERVENTIONS:
Drug: misoprostol — misoprostol 400mcg 12 hrs prior to procedure
  Other Names: Cytotec
  Arms: 2
Drug: vitamin B6 — Vitamin B6 50 mg orally 12 hrs prior to procedure
  Arms: 1

SUMMARY:
An endometrial biopsy involves a thin tube being passed through the cervix (opening of the uterus) to obtain a sample of the lining of the uterus. Sometimes there may be discomfort with this procedure especially if the cervix is not dilated or opened. Previous research has suggested that taking a drug called misoprostol may help the cervix to start to dilate or open. This study will see if misoprostol will help open the cervix for an endometrial biopsy, to lessen the discomfort and make the biopsy easier to perform.

ELIGIBILITY:
Inclusion Criteria:

* women 19 years and older
* planned endometrial biopsy

Exclusion Criteria:

* known hypersensitivity or allery to prostaglandins
* seizure disorder
* liver disease
* known abnormal liver function tests
* pregnancy

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2003-02; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
pain/discomfort of endometrial biopsy | during procedure

SECONDARY OUTCOMES:
ease of performing biopsy | during procedure
success of obtaining biopsy | during procedure
potential side effects | time study drug taken until procedure

CONTACTS AND LOCATIONS:
Overall Officials: Joan MG Crane, MD, Principal Investigator — Faculty, Discipline Obstetrics and Gynecology, Memorial University of Newfoundland
Locations (2):
- Canada (2):
  - Women's Health Centre, Eastern Health, St. John's, Newfoundland and Labrador
  - Obstetrics and Gynecology Associates, Dartmouth, Nova Scotia